CLINICAL TRIAL: NCT00004575
Title: Investigation of Miconazole as an Inhibitor of Endothelium-Derived Hyperpolarizing Factor
Brief Title: Effects of Miconazole on Blood Flow
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000077; 00-H-0077
Record Dates: First submitted 2000-02-17; First posted 2002-05-22 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-10

CONDITIONS: Healthy
Keywords: Endothelium; Vasodilation; Vascular Biology; Venous Occlusion Plethysmography
MeSH Terms: conditions — Aneurysm | interventions — Miconazole; omega-N-Methylarginine; Bradykinin

INTERVENTIONS:
Drug: Miconazole, L-NMMA, Bradykinin

SUMMARY:
This study will investigate the effect of the drug miconazole on blood vessel dilation. Miconazole stops production of EDHF, a substance that causes arteries to dilate. EDHF is produced by the cells that line blood vessels.

Normal volunteers between the ages of 21 to 60 may participate in this study. Candidates will be screened for eligibility with a medical history, physical examination, electrocardiogram and routine laboratory tests. Those enrolled will be injected with miconazole to study its effects on blood vessels.

Study participants will take three aspirin tablets. After administration of a local anesthetic, small tubes will be inserted through a needle into the artery and vein of the forearm. These will be used to measure blood pressure and to draw blood samples during the study. Forearm blood flow will be measured using pressure cuffs placed on the wrist and upper arm, and a strain gauge (a rubber band device) placed around the forearm. When the cuffs are inflated, blood will flow into the arm, stretching the strain gauge, and the flow measurement will be recorded.

Small doses of four drugs-bradykinin, sodium nitroprusside, miconazole, and LNMMA-will be given through the arterial catheter. Bradykinin stimulates the release of EDHF and can lower blood pressure. Sodium nitroprusside causes blood vessels to dilate and is used to treat high blood pressure and heart failure. Miconazole is commonly prescribed to treat various infections, including vaginal yeast infections, jock itch and athlete's foot. In much higher doses, it is used to treat fungal infections that have spread to the lungs, brain, kidneys, or bladder. LNMMA inhibits production of nitric oxide, another substance produced by the lining cells of blood vessels.

Blood flow will be measured throughout the study, which will last approximately 3 hours.

DETAILED DESCRIPTION:
The vascular endothelium synthesizes at least three potent vasodilator substances: nitric oxide (NO), prostacyclin and an endothelium-derived hyperpolarizing factor (EDHF). EDHF release is stimulated by receptor-dependent agonists such as acetylcholine and bradykinin (BK), and leads to hyperpolarization of the underlying smooth muscle cells presumably by opening Ca(2+)-activated K(+) channels. Indirect pharmacologic evidence suggests that EDHF is a cytochrome P450-derived arachidonic acid metabolite, presumably an epoxide.

Numerous inhibitors of EDHF have been defined in animal tissues. Of these, miconazole has proven to be safe when administered to humans as a topical and parenteral antifungal agent. At levels that are attained with routine clinical use, it has a rapid onset of action with high specificity of inhibition of EDHF in animal models. This study is designed to investigate the safety and efficacy of intra-arterial miconazole in inhibiting BK-mediated forearm vasodilation in normal volunteers.

ELIGIBILITY:
Healthy male or female volunteers (age 21-60 years).

No presence of intercurrent illness.

No current smoking (within previous 5 years).

No hypertension (greater than 140/90).

No diabetes.

No hypercholesterolemia (total cholesterol greater than 240 mg/dl).

No pregnancy or menopause.

No renal failure (creatinine greater than 1.4 mg/dl).

No allergies to miconazole, parabens, castor oil or aspirin.

No bleeding disorders.

No consumption of any medications during the last one week, including vitamins and unconventional medications.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 2000-02; Study Completion 2001-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Feletou M, Vanhoutte PM. Endothelium-derived hyperpolarizing factor. Clin Exp Pharmacol Physiol. 1996 Dec;23(12):1082-90. doi: 10.1111/j.1440-1681.1996.tb01174.x. PMID 8977164
- [Background] Furchgott RF, Vanhoutte PM. Endothelium-derived relaxing and contracting factors. FASEB J. 1989 Jul;3(9):2007-18. PMID 2545495
- [Background] Keef KD, Bowen SM. Effect of ACh on electrical and mechanical activity in guinea pig coronary arteries. Am J Physiol. 1989 Oct;257(4 Pt 2):H1096-103. doi: 10.1152/ajpheart.1989.257.4.H1096. PMID 2801972